CLINICAL TRIAL: NCT06268587
Title: A Before and After Study Studying the Impact of an Analgesia Protocol After Discharge From Outpatient Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Samalea Suarez Nicolas, MD, MD, Centre Hospitalier Universitaire de Liege
Other Study IDs: 2023/80
Record Dates: First submitted 2023-12-26; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Pain; Outpatient Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — argipressin, Asu(1,6)-

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control group: The control group is made up of patients, without age limit, who underwent an outpatient surgery from 01/09/19 to 28/02/20 inclusive and accepted post-operative monitoring by SMS. These patients leaves the hospital with instructions and prescriptions.
- experimental group: The experimental group is made up of patients, without age limit, who underwent an outpatient surgery procedure from 1/9/21 to 28/2/22 inclusive and accepted post-operative monitoring by SMS. The patients leaves the hospital with instructions, analgesics for a maximum of two days with detailed dosages and an explanatory booklet on postoperative pain.
  Interventions: Combination Product: Measure the impact of the home analgesia protocol on the proportion of patients with a VAS > 3/10 on day one and who did not take analgesics.

INTERVENTIONS:
Combination Product: Measure the impact of the home analgesia protocol on the proportion of patients with a VAS > 3/10 on day one and who did not take analgesics. — Measure the impact of the home analgesia protocol on the proportion of patients with a VAS > 3/10 on D+1 and who did not take analgesics. The protocol consists of providing the patient with instructions at the time of discharge, analgesics for a maximum of two days with dosages and an explanatory booklet on pain management
  Groups: experimental group

SUMMARY:
The goal of this before and after study is to measure the effectiveness of a home analgesia protocol after outpatient surgery in a tertiary hospital. The main question it aims to answer is:

- Measure the impact of the protocol on the proportion of patients with a VAS greater than 3/10 on day one and who did not take the analgesics.

The participants are divided into two groups. The control group leaves the hospital with instructions and prescriptions. The experimental group leaves the hospital with instructions, analgesics for a maximum of two days with detailed dosages and an explanatory booklet on postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* outpatient surgery
* no age limit
* accepted post-operative monitoring by text messages (SMS)

Exclusion Criteria:

* refusal of post-operative follow-up by text messages (SMS)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent outpatient surgery at the Liège university hospital center in Belgium
Sampling Method: Non-Probability Sample
Enrollment: 1423 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Measure the impact of the protocol on the proportion of patients with a pain greater than 3/10 on a Visual Analogue Scale at day one and who did not take the analgesics. | day 1
  Visual Analogue Scale = 0/10 : no pain Visual Analogue Scale = 10/10: maximal pain The patients receive a text message (SMS) on day 1 asking for their pain level between 1 and 10. They send the response via SMS. If the response is greater than 3/10, an SMS asks patients if they have taken their painkillers. If they took them, they say "taken". Otherwise, they are invited to take them and are contacted again 45 minutes later for a new evaluation.
  In the event of no response to the SMS or pain > 3/10 despite taking the prescribed painkillers, they are contacted by telephone.

SECONDARY OUTCOMES:
Measure the adequacy of post-op analgesics by measuring the proportion of patients with a Visual Analogue Scale < or = 3/10 on day one for each group | day 1
  Visual Analogue Scale = 0/10 : no pain Visual Analogue Scale = 10/10: maximal pain The patients receive a text message (SMS) on day 1 asking for their pain level between 1 and 10. They send the response via SMS. If the response is greater than 3/10, an SMS asks patients if they have taken their painkillers. If they took them, they say "taken". Otherwise, they are invited to take them and are contacted again 45 minutes later for a new evaluation.
  In the event of no response to the SMS or pain > 3/10 despite taking the prescribed painkillers, they are contacted by telephone.
Measure the impact of the protocol on the occurrence of nausea and vomiting on day one | day 1
  The patients receive a text message (SMS) on day 1 asking for their pain level between 1 and 10. The patients receive a text message (SMS) on day 1 asking if they suffer from nausea and vomiting. If the answer is no, they respond 0 to the SMS. If the answer is yes, they answer 1.
  In the event of no response to the SMS or the présence nausea and vomiting, they are contacted by telephone.
Measure the impact of the protocol on general satisfaction of stay in outpatient surgery on day 7 with a Visual Analogue Scale Satisfaction | day 7
  The patients receive a text message (SMS) on day 7 to know their satisfaction. A Visual Analogue Scale Satisfaction is used. A Visual Analogue Scale Satisfaction = 0: the worst experience. A Visual Analogue Scale Satisfaction = 10: the best experience

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Liège, Wallonia, Belgium